CLINICAL TRIAL: NCT05772754
Title: Molecular Pathways Involved in Cardiac Remodeling in Patients With Chronic Heart Failure With Preserved Ejection Fraction HFpEF by New Omics Technologies
Brief Title: Molecular Pathways Involved in Cardiac Remodeling in Patients With Chronic Heart Failure With Preserved Ejection Fraction by New Omics Technologies
Acronym: HFpEF
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Liuzzo Giovanna, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3671
Record Dates: First submitted 2023-02-14; First posted 2023-03-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Coronary Heart Disease
Keywords: molecular pathways; cardiac remodeling; coronary insufficiency
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: Partecipants with heart failure and pulmonary hypertension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chronic heart failure partecipants (Other): Patients in the Department of Cardiovascular Sciences with signs and symptoms of chronic heart failure, elevated natriuretic peptide levels, left atrial dilatation and/or left ventricular hypertrophy, ejection fraction greater than 50% on echocardiographic evaluation HFpEF
  Interventions: Genetic: study of molecular and protein pathways
- Chronic hert faiure and ejection fraction less than 40% at echocardiographic evaluation (Other): Patients admitted to the Department of Cardiovascular Sciences with signs and symptoms of chronic heart failure*, ejection fraction less than 40% at echocardiographic evaluation HFrEF
  Interventions: Genetic: study of molecular and protein pathways
- Partecipants with pulmonary hypertension (Other): Patients admitted with advanced HFpEF with development of pulmonary hypertension PH-HFpEF
  Interventions: Genetic: study of molecular and protein pathways
- Partecipants with advanced HFrEF (Other): Patients admitted with advanced HFrEF with development of pulmonary hypertension PH-HFrEF
  Interventions: Genetic: study of molecular and protein pathways
- Control Group (Other): 12 Controls (CTRL), recruited in the outpatient setting among subjects with cardiovascular disease, in the absence of heart failure
  Interventions: Genetic: study of molecular and protein pathways

INTERVENTIONS:
Genetic: study of molecular and protein pathways — 42 ml peripheral venous blood sample.
  Other Names: Analysis of protein profile; Genomics analysis

SUMMARY:
Heart failure with preserved ejection fraction nowadays affects about half of all patients with heart failure. In the general population, the prevalence of this subclass of heart failure (HFpEF, ed.) increases as the age of patients increases, especially in those over 65 years of age, and it has a significant gender. The study is to investigate the molecular pathways, predominantly protein patterns, involved in cardiac remodeling peculiar to heart failure with preserved ejection fraction (HFpEF) by comparing them with remodeling pathways and protein pattern alterations in patients with HFrEF. In addition, the study aims to identify molecular alterations that would allow early identification of the development of PH-HFpEF and PH-HFrEF, affecting the female gender more

DETAILED DESCRIPTION:
The study, placing itself within the framework of Translational Research, aims to gain a greater understanding of the different phenotypes of patients with HFpEF, to expand knowledge of the specific immune profile, and to identify new therapeutic targets for a heterogeneous clinical syndrome, to date lacking effective medical therapy. It is also proposed to find potential biomarkers with which to distinguish early between the two subclasses of decompensation and protein alterations related to the possible development of pulmonary hypertension in patients with HFpEF and HFrEF (PH-HFpEF and PH- HFrEF, respectively).

Patients who will take part in the study, following enrollment carried out on an inpatient or outpatient basis (being inpatients and control group subjects, respectively), will have follow-up visits at two times (at 1 month and at 6 months), in conjunction with regularly scheduled medical checkups, according to Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* heart failure patients

Exclusion Criteria:

* patients suffering from infectious diseases and serious infectious diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
The first aim of the study is to identify the protein expression to cardiac remodelling | 8 months
  Description of protein expression specific to cardiac remodelling underlying chronic heart failure with preserved ejection fraction, in relation to different patient comorbidities, so the primary objective will be to investigate the protein pathways at T0.

SECONDARY OUTCOMES:
Identify interaction variations between protein pathways | 6 months
  Identify the interaction networks between proteins using the protein set enrichment study. Using this software, identify the interaction circuits between the most highly expressed proteins, typical of each condition and shared between two clinical categories.
  This is important to identify the the change in the protein pathway with respect to baseline.
Analyze gene expression in patients with cronic heart failure | 6 months
  Identify the most highly expressed genes in the different clinical conditions under investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No